CLINICAL TRIAL: NCT04294719
Title: A Study of Cognitive Adaptation Training in Inpatient Forensic Environments
Acronym: finCAT
Status: Completed | Type: Observational
Sponsor: Centre for Addiction and Mental Health (Other)
Responsible Party: Principal Investigator, Sean Kidd, Chief of Psychology Division, Senior Scientist, Centre for Addiction and Mental Health
Other Study IDs: 115-2019
Record Dates: First submitted 2020-02-11; First posted 2020-03-04 (Actual); Results first posted 2023-01-26 (Actual); Last update posted 2023-01-26 (Actual); Status verified 2022-04

CONDITIONS: Schizophrenia
Keywords: Schizophrenia; Cognitive Adaptation Training; Forensic; Inpatient; Cognition; Environmental Supports
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Inpatient Clients: Have a chart diagnosis of a schizophrenia spectrum illness, capacity to consent or availability of a substitute decision-maker to consent with the assent of the participant and is residing on a CAMH inpatient forensic unit (general security)
  Interventions: Other: Cognitive Adaptation Training (CAT)

INTERVENTIONS:
Other: Cognitive Adaptation Training (CAT) — Cognitive Adaptation Training (CAT) is a standardized implementation of environmental supports for improving adaptive functioning including medication adherence, grooming, and daily activities in patients with schizophrenia. Environmental supports (signs, checklists) are manual-driven and grounded upon an assessment of neurocognitive function and behaviour. Assessment results yield one of six CAT classifications (Apathy/Poor Executive Functioning, Disinhibited/Poor EF, Mixed/Poor EF, Apathy/Fair EF, Disinhibited/Fair EF, Mixed/Fair EF).The goal will be to improve organization and self-care, modifying the intervention to be more relevant for an inpatient setting. Once an individual's CAT classification has been determined, strategies for specific functional problems are chosen from a series of tables. CAT interventions are maintained in the client's living space during weekly visits. CAT clinicians will encourage team members to assist with the reinforcement of CAT tools and strategies.

SUMMARY:
The proposed project will be a mixed-methods feasibility study of modified Cognitive Adaptation Training for an inpatient forensic mental health population (finCAT). Cognitive Adaptation Training (CAT) is an evidence-based compensatory cognitive intervention that focuses on improving functioning through the provision of environmental supports and cues. CAT is typically applied in outpatient care but has been successfully modified for inpatient service contexts in a Netherlands trial and at CAMH in previous pilots for both forensic and non-forensic inpatient populations.

DETAILED DESCRIPTION:
The proposed project will expand the investigators knowledge of the role of compensatory cognitive interventions for forensic inpatient populations with schizophrenia. Over the course of 6 months, the investigators will conduct a feasibility study of the delivery of a modified forensic inpatient version of Cognitive Adaptation Training. The objective of this single group study with pre-post and follow up assessments is to determine if preliminary outcomes and follow up findings support the feasibility of a modified version CAT within a forensic inpatient setting. Feasibility data will be used to inform (i) any necessary adjustments to the intervention, (ii) any necessary adjustments to the optimal time of study for outcomes to be observed, and (iii) to inform future trials with respect to anticipated recruitment and drop-out rates and optimal powering.

This study would be among the few examinations of CAT as an inpatient intervention to date, as well as the first to examine a modified cognitive adaptation training approach in both a North American and forensic inpatient setting, and would make a substantial contribution to the evidence-based intervention literature. This intervention will be referred to as forensic inpatient CAT or finCAT.

The questions for this project are:

1. Is finCAT feasible for forensic inpatient populations with a schizophrenia spectrum diagnosis? Based on preliminary work the investigators hypothesize that finCAT will prove acceptable to patients and inpatient staff and will demonstrate positive outcomes with respect to functioning and inpatient room organization.
2. What are the attitudes of inpatient forensic occupational therapists and clinical teams towards implementing finCAT on their units?

This study will expand on the preliminary work of the investigators at CAMH. The study will be implemented on four CAMH general security forensic inpatient units. There will be four weeks of CAT Clinician--delivered treatment focusing on two goal areas - room organization and personal hygiene, followed by two months of maintenance by CAT Unit Champions with pre, post, and two-month follow-up, as well as project-end evaluations. In the first four weeks, the investigators will conduct a trial of finCAT for two of the four inpatient general forensic units, followed by two months of finCAT maintenance with Unit CAT Champions supported by the CAT Clinician. This process would then be repeated on the remaining two general units at CAMH. Previous implementation of CAT has demonstrated gains within one-month; however, follow-up assessments were not conducted to determine if gains were maintained over time. While brief, this time period (i) reflects the intent of this study as a pilot test of feasibility and, (ii) aligns with this circumscribed version of CAT (as compared to the more comprehensive community version with broader outcome domains). Data will be collected from both primary participants (inpatients) and the clinical team.

ELIGIBILITY:
Inclusion Criteria:

1. A chart diagnosis of a schizophrenia spectrum illness.
2. Capacity to consent or availability of a substitute decision-maker to consent with the assent of the participant.
3. Participant residing on a CAMH inpatient forensic unit (general security)

Exclusion Criteria

1. High paranoia
2. Primary issue of hoarding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All participants will be recruited through CAMH Complex Care & Recovery inpatient forensic services.
Sampling Method: Non-Probability Sample
Enrollment: 24 (Actual)
Dates: Start 2019-12-12 (Actual); Primary Completion 2020-06-20 (Actual); Study Completion 2020-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sean Kidd, Principal Investigator — Centre for Addiction and Mental Health
Locations (1):
- Centre for Addiction and Mental Health, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No
Client-specific research data gathered as part of this study may be shared and provided to the paticipant's unit treatment team for client care. All client data gathered will be kept confidential within the participant's treatment team and the research project team. All other gathered data (i.e. staff data) will be kept de-identified, confidential, and anonymous.

REFERENCES:
- [Background] Alphs LD, Summerfelt A, Lann H, Muller RJ. The negative symptom assessment: a new instrument to assess negative symptoms of schizophrenia. Psychopharmacol Bull. 1989;25(2):159-63. No abstract available. PMID 2602512
- [Background] Aarons GA. Mental health provider attitudes toward adoption of evidence-based practice: the Evidence-Based Practice Attitude Scale (EBPAS). Ment Health Serv Res. 2004 Jun;6(2):61-74. doi: 10.1023/b:mhsr.0000024351.12294.65. PMID 15224451
- [Background] Brown S, Inskip H, Barraclough B. Causes of the excess mortality of schizophrenia. Br J Psychiatry. 2000 Sep;177:212-7. doi: 10.1192/bjp.177.3.212. PMID 11040880
- [Background] Chen S, Collins A, Anderson K, McKenzie K, Kidd S. Patient Characteristics, Length of Stay, and Functional Improvement for Schizophrenia Spectrum Disorders: A Population Study of Inpatient Care in Ontario 2005 to 2015. Can J Psychiatry. 2017 Dec;62(12):854-863. doi: 10.1177/0706743716680167. Epub 2016 Dec 14. PMID 29194005
- [Background] Draper ML, Stutes DS, Maples NJ, Velligan DI. Cognitive adaptation training for outpatients with schizophrenia. J Clin Psychol. 2009 Aug;65(8):842-53. doi: 10.1002/jclp.20612. PMID 19521972
- [Background] Frost, R. O., Steketee, G., Tolin, D. F., & Renaud, S. (2008). Development and validation of the clutter image rating. Journal of Psychopathology and Behavioral Assessment, 30(3), 193-203.
- [Background] Goeree R, Farahati F, Burke N, Blackhouse G, O'Reilly D, Pyne J, Tarride JE. The economic burden of schizophrenia in Canada in 2004. Curr Med Res Opin. 2005 Dec;21(12):2017-28. doi: 10.1185/030079905X75087. PMID 16368053
- [Background] Green MF. What are the functional consequences of neurocognitive deficits in schizophrenia? Am J Psychiatry. 1996 Mar;153(3):321-30. doi: 10.1176/ajp.153.3.321. PMID 8610818
- [Background] Harvey, P. D. (Ed.). (2013). Cognitive impairment in schizophrenia: Characteristics, assessment and treatment. Cambridge University Press.
- [Background] Hsieh HF, Shannon SE. Three approaches to qualitative content analysis. Qual Health Res. 2005 Nov;15(9):1277-88. doi: 10.1177/1049732305276687. PMID 16204405
- [Background] Kidd SA, Herman Y, Barbic S, Ganguli R, George TP, Hassan S, McKenzie K, Maples N, Velligan D. Testing a modification of cognitive adaptation training: streamlining the model for broader implementation. Schizophr Res. 2014 Jun;156(1):46-50. doi: 10.1016/j.schres.2014.03.026. Epub 2014 Apr 29. PMID 24794880
- [Background] Maples, N. J., & Velligan, D. I. (2008). Cognitive adaptation training: establishing environmental supports to bypass cognitive deficits and improve functional outcomes. American Journal of Psychiatric Rehabilitation, 11(2), 164-180.
- [Background] Rosen A, Hadzi-Pavlovic D, Parker G. The life skills profile: a measure assessing function and disability in schizophrenia. Schizophr Bull. 1989;15(2):325-37. doi: 10.1093/schbul/15.2.325. PMID 2749191
- [Background] Schalast N, Redies M, Collins M, Stacey J, Howells K. EssenCES, a short questionnaire for assessing the social climate of forensic psychiatric wards. Crim Behav Ment Health. 2008;18(1):49-58. doi: 10.1002/cbm.677. PMID 18229876
- [Background] Stiekema AP, Quee PJ, Dethmers M, van den Heuvel ER, Redmeijer JE, Rietberg K, Stant AD, Swart M, van Weeghel J, Aleman A, Velligan DI, Schoevers RA, Bruggeman R, van der Meer L. Effectiveness and cost-effectiveness of cognitive adaptation training as a nursing intervention in long-term residential patients with severe mental illness: study protocol for a randomized controlled trial. Trials. 2015 Feb 12;16:49. doi: 10.1186/s13063-015-0566-8. PMID 25887511
- [Background] Torrey WC, Drake RE, Dixon L, Burns BJ, Flynn L, Rush AJ, Clark RE, Klatzker D. Implementing evidence-based practices for persons with severe mental illnesses. Psychiatr Serv. 2001 Jan;52(1):45-50. doi: 10.1176/appi.ps.52.1.45. PMID 11141527
- [Background] van Dam, M., Stiekema, A., Islam, A., Swart, M., Redmeyer, J., Dethmers, M., ... & Bruggeman, R. (2017). SU15. Implementation of Cognitive Adaptation Training in a Hospital Setting: Facilitating and Hampering Factors. Schizophrenia bulletin, 43(Suppl 1), S166.
- [Background] van der Meer, L., Stiekema, A., van Dam, M., Swart, M., Redmeyer, J., Dethmers, M., ... & Pijnenborg, G. M. (2017). SU13. Cognitive Adaptation Training: Is It Effective as a Nursing Intervention in a Hospital Setting?. Schizophrenia bulletin, 43(Suppl 1), S165.
- [Background] Velligan, D. I., Mahurin, R. K., Eckert, S. L., Miller, A. L., & Bow-Thomas, C. C. (1997). Cognitive adaptation training: The use of compensatory strategies for inpatients and outpatients with schizophrenia. Schizophrenia Research, 1(24), 229.
- [Background] Velligan DI, Bow-Thomas CC, Huntzinger C, Ritch J, Ledbetter N, Prihoda TJ, Miller AL. Randomized controlled trial of the use of compensatory strategies to enhance adaptive functioning in outpatients with schizophrenia. Am J Psychiatry. 2000 Aug;157(8):1317-23. doi: 10.1176/appi.ajp.157.8.1317. PMID 10910797
- [Background] Velligan DI, Prihoda TJ, Ritch JL, Maples N, Bow-Thomas CC, Dassori A. A randomized single-blind pilot study of compensatory strategies in schizophrenia outpatients. Schizophr Bull. 2002;28(2):283-92. doi: 10.1093/oxfordjournals.schbul.a006938. PMID 12693434
- [Background] Velligan DI, Lam F, Ereshefsky L, Miller AL. Psychopharmacology: Perspectives on medication adherence and atypical antipsychotic medications. Psychiatr Serv. 2003 May;54(5):665-7. doi: 10.1176/appi.ps.54.5.665. No abstract available. PMID 12719495
- [Background] Velligan DI, Diamond PM, Mintz J, Maples N, Li X, Zeber J, Ereshefsky L, Lam YW, Castillo D, Miller AL. The use of individually tailored environmental supports to improve medication adherence and outcomes in schizophrenia. Schizophr Bull. 2008 May;34(3):483-93. doi: 10.1093/schbul/sbm111. Epub 2007 Oct 10. PMID 17932089
- [Background] Velligan DI, Diamond PM, Maples NJ, Mintz J, Li X, Glahn DC, Miller AL. Comparing the efficacy of interventions that use environmental supports to improve outcomes in patients with schizophrenia. Schizophr Res. 2008 Jul;102(1-3):312-9. doi: 10.1016/j.schres.2008.02.005. Epub 2008 Apr 18. PMID 18374542
- [Background] Williams, R.S. (June 2017). Occupational Therapists' Perspectives on Cognitive Adaptation Training. Poster presented at the Canadian Association of Occupational Therapists Conference, Charlottetown, PE, Canada.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Inpatient Clients
Started | 19
Completed | 18
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Inpatient Clients
Number analyzed (Participants) | 18
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.1 (10.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 17
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black | 12
  Caucasian | 6
Education [Count of Participants; unit: Participants]
  Less than High School | 2
  Some High School | 5
  High School | 5
  Some College | 2
  College Diploma | 2
  Some University | 1
  Undergraduate Degree | 1
Primary Diagnosis [Count of Participants; unit: Participants]
  Schizophrenia | 13
  Schizoaffective Disorder | 2
  Schizoaffective Bipolar | 3
Secondary Diagnosis [Count of Participants; unit: Participants]
  Antisocial Personality Disorder | 4
  Alcohol Dependence | 5
  Borderline Intelligence | 1
  Cannabis Use | 5
  Paraphilia Not Otherwise Specified | 1
  Substance Abuse | 1
  Substance Use | 4
  None | 1
Concurrent Diagnosis [Count of Participants; unit: Participants]
  Yes | 16
  No | 2
Dual Diagnosis [Count of Participants; unit: Participants]
  Attention Deficit Hyperactivity Disorder | 2
  ADHD and Intellectual Disability | 1
  Intellectual Disability | 2
  None | 13
Not Criminally Responsible/Unfit to Stand Trial Status [Count of Participants; unit: Participants]
  NCR | 18
  UST | 0
Violent Offense [Count of Participants; unit: Participants]
  Yes | 15
  No | 3
Approximate Age of First Episode [Mean (Standard Deviation); unit: years] | 21.3 (7.7)
Approximate Length of Illness (Years) [Mean (Standard Deviation); unit: years] | 16.8 (10.5)
Length of Stay (NCR Data-Treatment Start Date) [Mean (Standard Deviation); unit: days] | 2770.4 (2118.8)

OUTCOME MEASURES:

1. Primary Outcome: Clutter Image Rating Scale (CIRS) - Blind-rated
Description: Room organization will be measured by ratings on the Clutter Image Rating Scale (CIRS; Frost et al., 2008). The CIRS is a 9-picture visual analogue scale used to quantify and standardize the amount of clutter in 3 different living spaces (kitchen, living room, and bedroom). Min is 1 and Max is 9. Higher ratings indicate more clutter. For this project, only the bedroom rating scale will be utilized. The CIRS is used to measure the severity of clutter in compulsive hoarding. Before and after photos will be taken of each participant's room. These photos will be rated by 2 blinded student investigators with the mean rating taken.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Inpatient Clients
Number analyzed (Participants) | 18
score on a scale | 2.28 (.575)

2. Primary Outcome: Clutter Image Rating Scale (CIRS) - Blind-rated
Description: as for outcome 1
Time Frame: 4-Weeks Post-Intervention
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Inpatient Clients
Number analyzed (Participants) | 18
score on a scale | 1.56 (.616)

3. Primary Outcome: Clutter Image Rating Scale (CIRS) - Blind-rated
Description: as for outcome 1
Time Frame: 2-Month Follow-Up
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Inpatient Clients
Number analyzed (Participants) | 18
score on a scale | 1.44 (.511)

4. Primary Outcome: Clutter Image Rating Scale (CIRS) - Patient-rated
Description: as for outcome 1
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Inpatient Clients
Number analyzed (Participants) | 18
score on a scale | 1.94 (.80)

5. Primary Outcome: Clutter Image Rating Scale (CIRS) - Patient-rated
Description: as for outcome 1
Time Frame: 4-Weeks Post-Intervention
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Inpatient Clients
Number analyzed (Participants) | 18
score on a scale | 1.56 (.71)

6. Primary Outcome: Life Skills Profile (LSP) - Self-Care Subscale
Description: Personal hygiene will be measured by scores on the Life Skills Profile (LSP; Rosen, Hadzi-Pavlovic, & Parker, 1989). The LSP consists of 39 clinician-rated questions on a four-point scale and measures various aspects related to daily life activities: self-care; non-turbulence; social contact; communication; responsibility. For this project, only the self-care ratings from the full LSP-39 will be completed by service providers (items 10, 12, 13, 14, 15, 16, 23, 24, 26, and 30). While each item consists of 4 responses, the content of each response is different for each item. Overall, higher scores indicate better functioning. Max total score is 40. Min total score is 10. Current inpatient research on the use of CAT also uses this scale as a primary measure of the effectiveness of CAT. Scores will be obtained from the nursing staff not directly involved in the delivery of the finCAT intervention.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Inpatient Clients
Number analyzed (Participants) | 18
score on a scale | 23.56 (5.52)

7. Primary Outcome: Life Skills Profile (LSP) - Self-care Subscale
Description: as for outcome 6
Time Frame: 4-Weeks Post-Intervention
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Inpatient Clients
Number analyzed (Participants) | 18
score on a scale | 24.00 (5.64)

8. Primary Outcome: Life Skills Profile (LSP) - Self-care Subscale
Description: as for outcome 6
Time Frame: 2-Month Follow-Up
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Inpatient Clients
Number analyzed (Participants) | 18
score on a scale | 24.61 (4.79)

9. Primary Outcome: Goal Attainment Scaling (GAS) - Goal 1
Description: Goal Attainment Scaling (GAS) will be employed as a sensitive measure of progress on individually defined goals. Goal attainment scaling involves the setting of 3-5 goals, each operationalized on a 5-point scale. Min is -2. Max is 2. Higher scores indicate greater attainment of the goal. Goals are individualized to the client and assessment of progress is determined through consensus of the clinician and case manager.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Inpatient Clients
Number analyzed (Participants) | 18
score on a scale | -1.00 (.000)

10. Primary Outcome: Goal Attainment Scaling (GAS) - Goal 1
Description: as for outcome 9
Time Frame: 4-Week Post-Intervention
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Inpatient Clients
Number analyzed (Participants) | 18
score on a scale | 1.06 (.984)

11. Primary Outcome: Goal Attainment Scaling (GAS) - Goal 1
Description: as for outcome 9
Time Frame: 2-Month Follow-Up
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Inpatient Clients
Number analyzed (Participants) | 18
score on a scale | 0.81 (.889)

12. Primary Outcome: Goal Attainment Scaling (GAS) - Goal 2
Description: as for outcome 9
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Inpatient Clients
Number analyzed (Participants) | 18
score on a scale | -1.00 (.000)

13. Primary Outcome: Goal Attainment Scaling (GAS) - Goal 2
Description: as for outcome 9
Time Frame: 4-Week Post-Intervention
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Inpatient Clients
Number analyzed (Participants) | 18
score on a scale | 1.11 (1.13)

14. Primary Outcome: Goal Attainment Scaling (GAS) - Goal 2
Description: as for outcome 9
Time Frame: 2-Month Follow-Up
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Inpatient Clients
Number analyzed (Participants) | 18
score on a scale | 0.78 (.878)

15. Secondary Outcome: Evidence-Based Practice Attitude Scale (EBPAS)
Description: The attitudes of the team members towards finCAT will be measured using the Evidence-Based Practice Attitude Scale (EPBAS; Aarons, 2004) adapted to specifically target attitudes towards CAT. The EPBAS is a self-report questionnaire consisting of 36 items measured on a 5-point Likert scale ranging from 0 ('Not at all') to 4 ('To a very great extent') and consists of 12 subscales. Maximum is 4. Minimum is 0. Higher scores indicate a more open attitude towards new types of therapy, interventions or treatments including manualized therapy.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Allied Health Clinicians: Occupational therapists, behaviour therapists, recreation therapists, & social workers recruited and trained to act as unit-based CAT Point People, as well as 12 nurses and 2 managers from participating units.
- Nurses: Nursing staff working on the units where finCAT was administered.
Arm/Group | Allied Health Clinicians | Nurses
Number analyzed (Participants) | 15 | 12
score on a scale | 3.15 (.35) | 2.83 (.70)

16. Secondary Outcome: Evidence-Based Practice Attitude Scale (EBPAS)
Description: as for outcome 15
Time Frame: 2-Month Follow-Up
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Allied Health Clinicians | Nurses
Number analyzed (Participants) | 15 | 12
score on a scale | 3.22 (.24) | 2.92 (.55)

17. Secondary Outcome: Essen Climate Evaluation Schema (Essen CES)
Description: The therapeutic alliance on the unit will be measured by clinician and client ratings on the Essen Climate Evaluation Schema (Essen CES; Schalast et al., 2008). The Essen CES is a 15-item questionnaire measured on a 5-point Likert scale ranging from 'Not at all' to 'Very Much' and consists of three subscales: (1) Patient's Cohesion, (2) Experienced Safety, and (3) Therapeutic Hold. For this study, client and clinician ratings on the Therapeutic Hold and Experienced safety subscales will be collected. For each sub-scale, the max is 20 and minimum is 0. Higher scores indicate greater experienced safety and therapeutic hold.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Inpatient Clients | Allied Health Clinicians | Nurses
Number analyzed (Participants) | 18 | 15 | 12
score on a scale
  Experienced Safety | 13.46 (3.60) | 10.94 (3.28) | 10.67 (4.55)
  Therapeutic Hold | 12.85 (4.36) | 15.19 (3.39) | 14.67 (2.94)

18. Secondary Outcome: Essen Climate Evaluation Schema (Essen CES)
Description: as for outcome 17
Time Frame: 2-Month Follow-Up
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Inpatient Clients | Allied Health Clinicians | Nurses
Number analyzed (Participants) | 18 | 15 | 12
score on a scale
  Experienced Safety | 13.15 (3.56) | 11.06 (3.17) | 12.17 (2.48)
  Therapeutic Hold | 12.77 (4.68) | 15.25 (2.89) | 15.83 (1.17)

19. Secondary Outcome: Qualitative Care Provider Attitudes
Description: The attitudes of the team members towards finCAT will also be measured using a qualitative feedback form created for this study. Questions will target attitudes towards finCAT, perceptions of the impact of finCAT, and perceptions of team tension or conflict arising or abating during the implementation of finCAT. Small focus groups with healthcare providers will be facilitated by student investigators. Interviews will be audio-recorded and transcribed verbatim.
Time Frame: 2 months after month of service implementation
Reporting Status: Not Posted

20. Secondary Outcome: Qualitative Participant Attitudes
Description: The attitudes of the participants towards finCAT will also be measured using a qualitative feedback form created for this study. Questions will target attitudes towards finCAT, perceptions of the impact of finCAT. Individual interviews with interested clients will be facilitated by student investigators. Interviews will be audio-recorded and transcribed verbatim.
Time Frame: 2 months after month of service implementation
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Inpatient Clients
All-Cause Mortality (participants affected / at risk) | 0/18
Serious Adverse Events (participants affected / at risk) | 0/18
Other Adverse Events (participants affected / at risk) | 0/18

LIMITATIONS AND CAVEATS:
Sample size is lower than what would be ideal for feasibility trials and leave analyses under-powered to a degree. Lack of a control group limiting generalizability. Due to the COVID-19 pandemic, adaptations were made to the study design to accommodate procedural changes and patient safety.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-11-18): https://cdn.clinicaltrials.gov/large-docs/19/NCT04294719/Prot_SAP_000.pdf
  • Informed Consent Form (2019-11-01): https://cdn.clinicaltrials.gov/large-docs/19/NCT04294719/ICF_001.pdf